CLINICAL TRIAL: NCT02800005
Title: Effect of Obesity on Surgical Outcomes and Survival for Gastric Cancer Patients: a Single Center Prospective Cohort Study
Brief Title: Effect of Obesity on Surgical Outcomes and Survival for Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jian-Kun Hu (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Jian-Kun Hu, M.D. Ph.D., West China Hospital
Organization: West China Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: WCH-GC-04
Record Dates: First submitted 2016-02-24; First posted 2016-06-15 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Obesity; Gastric Cancer
Keywords: gastric cancer; gastrectomy; laparotomy; surgical outcome; survival; abdominal fat area; Body Mass Index
MeSH Terms: conditions — Obesity; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMI group (Successive patients) (Other): All successive patients meeting the including criteria and signed the informed consent will be measured BMI and the data will be recorded in the prospective database. The formula for BMI is weight in kilograms divided by height in meters squared (kg/m2). the normal range is usually considered to be 18.5 to 24.9, with less than 18.5 considered underweight, more than 25.0 considered overweight and above 30.0 obese. Investigators declare that there exists no conflicts of interest.
  Interventions: Other: BMI group (successive patients)
- AFA group(Successive patients) (Experimental): All successive patients meeting the including criteria and signed the informed consent will be measured BMI and the data will be recorded in the prospective database. The abdominal fat area at the umbilical level was measured using a CT scanner(sango Mount Monitor Wireless Panel; Siemens , Munich, Germany) while the examinee was in a supine position and estimated using a Volume software (fat Pointer; Siemens , Munich, Germany). The imaging conditions were 120 kilovolt and 50 milliampere, using a 5-mm-thick slice.The areas covered by visceral fat software calculated from pixels with densities ranging from-190 to -30 hounsfield unit. No contrast agent is needed. Patients in the AFA group will be also measured by BMI. Investigators declare that there exists no conflicts of interest.
  Interventions: Device: AFA group (successive patients); Other: BMI group (successive patients)

INTERVENTIONS:
Device: AFA group (successive patients) — The abdominal fat area at the umbilical level was measured using a CT scanner(sango Mount Monitor Wireless Panel; Siemens , Munich, Germany) while the examinee was in a supine position and estimated using a Volume software (fat Pointer; Siemens , Munich, Germany). The imaging conditions were 120 kilovolt and 50 milliampere, using a 5-mm-thick slice.The areas covered by visceral fat software calculated from pixels with densities ranging from-190 to -30 hounsfield unit . No contrast agent is needed.
  Arms: AFA group(Successive patients)
Other: BMI group (successive patients) — The formula for BMI is weight in kilograms divided by height in meters squared (kg/m2). the normal range is usually considered to be 18.5 to 24.9, with less than 18.5 considered underweight, more than 25.0 considered overweight and above 30.0 obese.

SUMMARY:
As the number of obesity continues to increase, surgical oncologist pay more attention to the effect of obesity on surgical outcomes and survival of digestive systemin cancers. Body mass index(BMI) is one of the most widely used measurements of obesity. Abdominal fat area (AFA) calculated by computed tomography is popular because of its validity of fat distribution. There is still no consensus which of BMI and AFA could be the more effective measurement and more accurate to evaluate effect of obesity on surgical outcomes and survival. Gastric cancer is one of the most common digestive system cancers, and gastrectomy is the primary therapeutic options.It is important to compare the different measurements(BMI or AFA) to assess obesity and effect on surgical outcome and survival for gastric cancer patients.

DETAILED DESCRIPTION:
Standard operation procedure（SOP）

1. Preoperative evaluation Patients satisfied with inclusion/exclusion criteria will be informed to join in the clinical study and signature the inform consent.
2. Procedures: The surgical treatments is adopted total or subtotal gastrectomy according to the Japanese Gastric Cancer treatments guidelines, 2010, Version 3.
3. Postoperative recovery: Postoperative recovery period need to collect those relevant parameters of all the patients. All the relevant parameters had definitely definition in the Case Report Form of this study which included the preoperative, intraoperative and postoperative clinicopathologic characteristics.
4. Follow-up: Follow-up will last to 5-year of the postoperative period. The postoperative complications is graded by the clavian-dildo classification. The postoperative complications and quality of life (change of AFA,performance status, recurrence and overall survival)are the focus of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative endoscopy and biopsy confirmed gastric adenocarcinoma, and predictively feasible of conventional open total gastrectomy or subtotal gastrectomy;
2. Predictively resectable diseases, of preoperative staging Japanese Gastric Cancer Association 14th Edition clinical T1N0M0-T4aN+M0;
3. Age：≤75 years, or ≥18 years;
4. Without serious disease and malignance disease;
5. Without histories of abdominal surgery;
6. World Health Organization performance score ≤2, American Society of Anesthesiologists score ≤3;
7. No limit to sexual and race;
8. Informed consent required;
9. Obesity is defined as BMI≧30kg/m2 or preoperative AFA≧100cm2/cm.

Exclusion Criteria:

1. Patients with other severe complications cannot tolerate surgery: such as severe heart and lung diseases, heart function below clinical stage 2, uncontrollable hypertension, pulmonary infection, moderate to severe chronic obstructive pulmonary disease, chronic bronchitis, severe diabetes and / or renal insufficiency, severe hepatitis and / or function below the rank of CHILD B grade, and severe malnutrition, etc;
2. Patients treated with neoadjuvant chemotherapy or radiation therapy which might affect the efficacy observation;
3. Severity mental diseases;
4. Primary lesion cannot be resected in the pattern of transabdominal gastrectomy, but for Whipple's procedure, or with a transthoracic approach surgery;
5. After signature the Clinical trial agreement, patients and their agent will quit the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 30-day of postoperative duration
  The criteria of postoperative complications in the BMI group and AFA group both adopt the definition of The clavian-dildo classification of surgical complications: five-year experience. Ann Surg. 2009;250 (2):187-96.Postoperative complications in Grade 1 were classified as minor complications, while complications in Grade 2 to 5 were classified as major complications.

SECONDARY OUTCOMES:
Change of the postoperative BMI | 5-year of postoperative duration.
  The body weight(kilograms) and height(meters) change of all enrollment after 5-year postoperative duration were measured to get the change of BMI.The formula for BMI is weight in kilograms divided by height in meters squared (kg/m2). The change of BMI was compared between preoperation and 5-year postoperative duration.
Change of the postoperative AFA | 5-year of postoperative duration
  AFA of all enrollment after 5-year postoperative duration were measured by CT. The AFA at the umbilical level was measured using a CT scanner (sango Mount Monitor Wireless Panel; Siemens , Munich, Germany) while the examinee was in a supine position and estimated using a Volume software (fat Pointer; Siemens , Munich, Germany). The imaging conditions were 120 kilovolt and 50 milliampere, using a 5-mm-thick slice. The areas covered by visceral fat software calculated from pixels with densities ranging from-190 to -30 hounsfield unit. The change of AFA was compared between preoperation and 5-year postoperative duration.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Kun Hu, M.D.Ph.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang SJ, Li HR, Zhang WH, Liu K, Zhang DY, Sun LF, Chen XL, Zhao LY, Chen XZ, Yang K, Chen ZX, Zhou ZG, Hu JK. Visceral Fat Area (VFA) Superior to BMI for Predicting Postoperative Complications After Radical Gastrectomy: a Prospective Cohort Study. J Gastrointest Surg. 2020 Jun;24(6):1298-1306. doi: 10.1007/s11605-019-04259-0. Epub 2019 Jun 3. PMID 31161593